CLINICAL TRIAL: NCT03995914
Title: Impact of Depression on 1-year Major Adverse Events in Patients Aged 75 or Older Who Undergo Transcatheter Aortic Valve Implantation (TAVIDEP)
Brief Title: Depression and Major Adverse Events in Older Patients Who Undergo a Transcatheter Aortic Valve Implantation
Acronym: TAVIDEP
Status: Withdrawn | Type: Observational
Why Stopped: Reclassification by Ethics Committee
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0295
Record Dates: First submitted 2019-06-13; First posted 2019-06-24 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-06

CONDITIONS: Depression; Aortic Stenosis
Keywords: MACCEs; Major cardiac and cerebrovascular events; TAVI; Older
MeSH Terms: conditions — Depression; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Depression, screened using the Geriatric Depression Scale (GDS) Short Form, has recently been found to be associated with a 3-fold increase in 1-year mortality after aortic valve replacement (AVR) in patients aged 70 or older. The main objective of the study is to evaluate whether the 1-year incidence of major adverse cardiac and cerebrovascular events (MACCEs), evaluated according to the valve academic research consortium 2 (VARC-2 criteria), in patients aged 75 or older who undergo a transcatheter aortic valve implantation (TAVI), should be similar in patients with depression systematically screened (using the 15-item GDS score), confirmed, and handled by a psychiatrist, and in patients without depression detected, after adjusting for frailty criteria and comorbidities.

DETAILED DESCRIPTION:
* Setting: the University hospital of Montpellier and the Perpignan hospital (France)
* Study population: 300 patients undergoing a TAVI, recruited over a 2-year period and followed for 12 months.
* Measurements at baseline: depression systematically screened by the 15-item Geriatric Depression Scale before TAVI. If the score is 4 or higher, patients will be evaluated by a psychiatrist and the patient will be treated according to current guidelines. Other possible confounders of the relationship between depression and poor outcomes: age; Fried's frailty phenotype; short physical performance battery; comorbidities; disability in the activities of daily living (ADL) and instrumental activities of daily living (IADL); cognitive function (Mini Mental State Examination; Clock Test score; Montreal cognitive assessment).
* Measurements (by telephone): 30 days after TAVI: MACCEs and hospitalization stay duration; 6 and 12 months after TAVI: MACCEs, 15-item GDS, ADL and IADL, new medical problem since the last visit, hospital admission, death, compliance and adverse effects of antidepressant drugs if applicable.

In case of withdrawal, the investigator will perform all examinations scheduled for the final study visit, which includes recording of AEs. In any case, the patient will be treated in accordance with standard care in the Montpellier and Perpignan centers.

Our hypothesis is that 40% of patients aged 75 or older will meet the criteria for depression (1-2), and that the 12-month incidence of MACCEs will be of 25% in patients without depression and of 50% in patients with depression. Our assumption is that the treatment of depression will reduce by 50% the incidence of MACCEs, to reach comparable incidence (relative difference of 10% or less) as the incidence observed in patients without depression.

To test this hypothesis, the number of patients with depression is 110 and the number of patients without depression is 165 (Total: 275 patients) to have a power of 90%. Considering a loss to follow-up rate of 10%, 300 patients will be included in the present study.

-Population analysis : The data will be entered into an eCRF (Ennov clinical) allowing consistencies control and remote monitoring. The data will also be validated on site from the source data by the TEC of the study. All included subjects will be taken into account in the description of the population. Data will be analyzed under the responsibility of Marie-Christine PICOT (Epidemiology and clinical research unit of the Montpellier University Hospital) with SAS software version 9 (SAS Institute, Cary, N.C.).

The statistical analysis plan (SAP), covering all the analyses to be performed on all data, will be written before database lock. For all collected variables, descriptive statistics will be calculated according to the level of measurement. For metric variables, a check whether the data can be assumed normally distributed will be first conducted. For normally distributed variables, mean and standard deviation will be calculated. For skewed variables, median and range will be used. In case of categorical variables group proportions and contingency tables will be prepared.

A comparison of baseline parameters between patients with and without depression (age, gender, number of drugs taken, Fried's and Rockwood's frailty criteria, SPPB, TUG, HRQOL, ADL, IADL, MMSE, Clock-Drawing test, MOCA; lives alone or not) will be conducted.

The incidence of MACCEs and other endpoints (mortality, hospitalization and nursing home admission rate, ADL, IADL score) at 6 and 12 months after TAVI will be compared between patients screened and treated for depression and in patients without depression. All analyses will be performed before and after adjustment for parameters distinguishing patients with confirmed depression and without depression at baseline.

The efficacy of the treatment of depression started by the psychiatrist will be assessed by comparing the 15item GDS, CES-D, Lille Apathy rating scale, HRQOL at baseline and at 6 and 12 months. The AE of antidepressant drugs will be described, such as the rate of withdrawal.

If the incidence of MACCEs and other outcomes is comparable in both groups of patients, the present study will provide preliminary results in order to conduct a randomized control trial to demonstrate that the systematic screening of depression and its treatment can reduce the incidence of MACCEs in patients aged 75 or older who undergo a TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years or older
* Patients eligible for TAVI and for study inclusion after a consensus decision of a multidisciplinary team including at least an interventional cardiologist, a cardiothoracic surgeon, a geriatrician, and an anesthetist.
* Subjects able to attend all scheduled visits and to comply with all trial procedures
* Subjects covered by public health insurance
* Signed informed

Exclusion Criteria:

* Subject unable to read or/and write
* Patients with emergency procedure, clinical instability (defined as unstable vital signs or refractory ongoing symptoms, acute decompensated heart failure)
* Patients with severe neuropsychiatric impairment
* Planned longer stay outside the region that prevents compliance with the visit plan
* Subject who are in a dependency or employment with the sponsor or the investigator
* Participation in another clinical trial within the last 4 weeks before the screening date

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 75 years or older, admitted for TAVI for severe and symptomatic aortic stenosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Incidence of MACCEs | 1 year
  Incidence of MACCEs (VARC-2 criteria) 12 months after a TAVI in patients aged 75 or older with or without depression screened using 15-item GDS and confirmed and handled by a psychiatrist.

SECONDARY OUTCOMES:
Number of Incidence of MACCEs | 1 and 6 months
  MACCEs (VARC-2 criteria) 1 and 6 months after a TAVI in patients aged 75 or older with or without depression screened using 15-item GDS and confirmed and handled by a psychiatrist
Number of Death | 6 and 12 months
  Death change 6 and 12 months after a TAVI in patients aged 75 or older with or without depression screened using 15-item GDS and confirmed and handled by a psychiatrist.
Number of hospitalization | 6 and 12 months
  Hospitalization change 6 and 12 months after a TAVI in patients aged 75 or older with or without depression screened using 15-item GDS and confirmed and handled by a psychiatrist.
Katz Index of Independence in Activities of Daily Living | 6 and 12 months
  Bathing, Dressing, toileting, Transferring, Continence, Feeding. SCORING: 6 = High (patient independent for activities of daily living) 0 = Low (patient very dependent for activities of daily living)
The Lawton Instrumental Activities of Daily Living (IADL) Scale | 6 and 12 months
  Ability to Use Telephone, Shopping, Food Preparation, Housekeeping, Laundry, Ability to Handle Finances. SCORING: 8 = High (patient independent for instrumental activities of daily living) 0 = Low (patient very dependent for instrumental activities of daily living)
Rate of depression | 1, 6 and 12 months
  Rate of depression confirmed by a psychiatrist when a depression has been screened using the 15-item Geriatric Depression Scale (Are you basically satisfied with your life, Have you dropped many of your activities and interests, Do you feel that your life is empty, Do you often get bored, Are you in good spirits most of the time, Are you afraid that something bad is going to happen to you, Do you feel happy most of the time, Do you often feel helpless, Do you prefer to stay at home, rather than going out and doing new things, Do you feel you have more problems with memory than most, Do you think it is wonderful to be alive now, Do you feel pretty worthless the way you are now, Do you feel full of energy, Do you feel that your situation is hopeless, Do you think that most people are better off than you are; Score : > 5 points is suggestive of depression, ≥ 10 points is almost always indicative of depression, > 5 points should warrant a follow-up comprehensive assessment)
Compliance of anti-depressant drugs prescribed | 1, 6 and 12 months
  Compliance of anti-depressant drugs prescribed in patients diagnosed with depression by a psychiatrist after a systematic. Center for Epidemiologic Studies- Depression scale. 20 questions with a value of 0, 1, 2 or 3 depending on the response (I was bothered by things that usually don't bother me, I did not feel like eating; my appetite wasn poor, I felt that I could not shake off the blues even with help from my family or friends, I felt I was just as good as other people, I had trouble keeping my mind on what I was doing, I felt depressed, I felt that everything I did was an effort, I felt hopeful about the future, I thought my life had been a failure, I felt fearful, My sleep was restless, I was happy, I talked less than usual, I felt lonely, People were unfriendly, I enjoyed life, I had crying spells, I felt sad, I felt that people disliked me, I could not get "going. Score : Less than 15, 15-21, Mild to Moderate Depression, Over 21, Possibility of Major Depression)
Effects of anti-depressant drugs prescribed on the Health | 1, 6 and 12 months
  Effects of anti-depressant drugs prescribed in patients diagnosed with depression by a psychiatrist after a systematic. The Short Form (36) Health Survey (a 36-item, patient-reported survey of patient health).
  vitality eight scaled scores (disability, physical functioning, bodily pain, general health perceptions ; physical role functioning ;emotional role functioning ; social role functioning ; mental health, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: hubert Blain, MD, PhD, Principal Investigator — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Result] Drudi LM, Ades M, Turkdogan S, Huynh C, Lauck S, Webb JG, Piazza N, Martucci G, Langlois Y, Perrault LP, Asgar AW, Labinaz M, Lamy A, Noiseux N, Peterson MD, Arora RC, Lindman BR, Bendayan M, Mancini R, Trnkus A, Kim DH, Popma JJ, Afilalo J. Association of Depression With Mortality in Older Adults Undergoing Transcatheter or Surgical Aortic Valve Replacement. JAMA Cardiol. 2018 Mar 1;3(3):191-197. doi: 10.1001/jamacardio.2017.5064. PMID 29344620